CLINICAL TRIAL: NCT00920621
Title: Randomized Trial: Maternal Vitamin D Supplementation to Prevent Childhood Asthma (VDAART)
Acronym: VDAART
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Scott T. Weiss, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 655; 5U01HL091528-03 (NIH); HL091528-01A1
Record Dates: First submitted 2009-06-11; First posted 2009-06-15 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Asthma
Keywords: Asthma; Vitamin D; Randomized Control Trial
MeSH Terms: conditions — Asthma | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D treatment (Experimental): vitamin D treatment plus prenatal multivitamins
  Interventions: Dietary Supplement: Vitamin D 3 cholecalciferol; Dietary Supplement: Vitamin D3
- placebo (Placebo Comparator): placebo plus prenatal multivitamins
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D 3 cholecalciferol — Dosage form oral Dosage 4000IU Vitamin D 3 cholecalciferol
  Other Names: vitamin D; vitamin D3; cholecalciferol
  Arms: Vitamin D treatment
Dietary Supplement: Vitamin D3 — 4000 IU of vitamin D3 administered orally once a day during pregnancy

SUMMARY:
Vitamin D supplementation given to pregnant women will prevent asthma in their offspring and children.

DETAILED DESCRIPTION:
Asthma is one of the leading causes of morbidity in children with 60% of all cases diagnosed by age 3. Thus, finding factors that can lead to prevention of this disease would be of great public health importance. Vitamin D deficiency is highly prevalent among pregnant women, and thus, represents a potentially modifiable factor for the prevention of disease. Due to the effect of vitamin D in modulating immune responses, we believe that vitamin D deficiency in pregnant mothers leads to faulty immune system development in the neonate, predisposing them to asthma and allergy. We have observational data from two independent birth cohort studies that higher maternal intakes of vitamin D during pregnancy are each independently associated with a 50% reduction in risk for recurrent wheezing and asthma in 3- and 5-yr old children. However, in order to recommend this as a universal treatment to prevent asthma, a randomized, controlled, clinical trial is necessary. Therefore, we propose a two arm, double-blind, placebo controlled, randomized, clinical trial of Vitamin D, to determine whether higher vitamin D intake and levels in the pregnant mother will prevent asthma and allergy in the child at age 3. We will identify pregnant women who have asthma or allergies or whose partner has asthma or allergies, from obstetric clinics in the three clinical centers participating in this trial. We will recruit 870 pregnant women during the first trimester of pregnancy and randomize them to one of two treatment arms of a 4-year clinical trial: 4000 IU of Vitamin D in addition to usual prenatal vitamins, n=435; and usual prenatal vitamins alone, n=435. Our primary specific aim is to determine whether adequate vitamin D supplementation in the pregnant mother is associated with reduced incidence of asthma in the child during the first 3 years of life. The sub-aims of the study will include (1) To determine whether adequate vitamin D supplementation in the pregnant mother is associated with reduced secondary outcomes in the child of (a) allergic sensitization, (b) doctor's diagnosis of eczema and (c) lower respiratory tract infections during the first 3 years of life; and (2) To determine whether adequate vitamin D supplementation in the pregnant mother is associated with improved vitamin D status in the mothers and their offspring through measurement of 25(OH)D levels in maternal plasma, cord blood, and children's blood at 1 and 3 yrs of age and (3)To determine whether sufficient vitamin D supplementation in the pregnant mother is associated with reduced incidence of preterm birth (birth <37 weeks gestation), preeclampsia, gestational hypertension, and/or Hemolytic anemia, Elevated Liver enzymes, Low Platelet count (HELLP syndrome) (PB/PE) compared to a usual care control group in VDAART.

VDAART Analysis Plan (Addendum to Protocol)

All analyses of primary and secondary outcomes stated in the VDAART Protocol will be performed using the intent-to-treat (ITT) paradigm, unless specifically stated.

I. Definition of outcomes.

A. Asthma and recurrent wheezing. The primary outcome of the trial will be development of a doctor's diagnosis of asthma and/or recurrent wheeze. While asthma is acknowledged to have its roots in early life, making a definite diagnosis is difficult until the child is older, and wheezing illnesses may be precursors of an asthma diagnosis. Thus, we will have a composite definition for the primary outcome.

* Asthma will be defined as a parent's report of physician's diagnosis at any time during the first three years of life, based on questionnaire responses. For time-to-event analyses, the time of incident asthma will be determined by the time of first positive questionnaire response.
* Recurrent wheezing will be defined as at least one report of wheezing in the third year of life plus any report of wheezing in any of the first two years of life.

Recognizing that wheezing symptoms may be modified by medication use, variable age of onset, and other variables, the following will be included in the composite outcome:

* children who had at least one wheezing episode (during the 1st 2 years of life), plus an asthma controller medication (defined as steroid inhalers or nebulizers OR steroid pills or liquids OR leukotriene modifiers) in the third year
* children who did not report any wheezing in the first 2 years but who report 2 separate episodes of wheezing in the third year OR are on controller medication (defined as above) on at least 2 separate reports in the third year OR at least 1 report of wheezing and at least 1 separate report of controller medication use in the third year

For recurrent wheezing (and the other wheezing phenotypes), the time of incident recurrent wheezing will be determined by the time of first report of wheezing, for time-to-event analyses. In the event that the child meets the definition based solely on the use of controller medication, the first report of use of this controller medication will be used to determine the time of onset of wheezing for time-to-event analyses.

For these outcomes, because the questions were asked every 3 months, and recognizing that missing questionnaires occurred, event times will be treated as interval-censored.

B. Eczema. Eczema will be defined as a positive response to parent's report of physician's diagnosis at any time during the first three years of life based on the questionnaire responses.

C. Lower respiratory tract infections (LRI). Lower respiratory tract infections (LRIs) will be defined based on parental responses to questionnaires. LRIs will be defined as a parental report of a physician's diagnosis of pneumonia, bronchiolitis, bronchitis, or croup (laryngotracheobronchitis). LRIs may occur multiple times over a three-year period in a child. Information on repeated episodes of LRI will be employed for rate estimation and comparison.

D. Total and specific IgE. Total and specific serum IgE will be measured from cord blood samples, and from year 3 samples from the children. Total IgE will be analyzed as a continuous outcome. Sensitization will be defined as any specific IgE ≥ 0.35 IU.

II. Secondary Analyses.

A. Analyses based on levels. Secondary analyses using baseline and follow-up maternal 25OHD levels will be performed. We will investigate the effect of baseline and follow-up maternal levels separately on the development of primary and secondary outcomes in the trial. Additionally, we will categorize mothers into categories based on joint baseline and follow-up levels. Mothers who have baseline levels and follow-up levels ≥ 40 mg/dl will be categorized in the HI-HI group; those who have baseline levels and follow-up levels < 40 mg/dl will be categorized in the LO-LO group; mothers who do not meet these definitions will be categorized either in the HI-LO or LO-HI groups based on their baseline and follow-up levels.

B. We also performed metabolomics on the children at age 1 and 3 and eventually age 6. We are assessing the association with vitamin D, asthma, and other phenotypes such as food allergies, IgE, and lung function with metabolites and genetic variants.

C. As an ancillary study, we have collected stool samples from the mothers in the 3rd trimester, and samples from the infants and children at 3-6 months, 1 year, and 3 years. We will sequence the stool samples for the microbiome, and we will assess the effects of the early life microbiome on the development of asthma, allergies (including food allergies and sensitization), growth and development, and obesity.

D. In a secondary analyses, we will determine the effect of 17q21 genotype on the efficacy of vitamin D supplementation in the prevention of asthma/wheeze. We will compute hazard ratios for the reduction in asthma/wheeze risk associated with prenatal supplementation, stratified by rs12936231. rs12936231 is a functional SNP influencing expression of ORMDL3, and given the role of ORMDL3 as a key sphingolipid biosynthesis regulator, we will subsequently investigate the relative abundance of sphingolipids between those in the vitamin D Intervention arm and those in the placebo group, stratified by 17q21 genotype. Relative abundance is quantified by normalizing the peak area of a metabolite to the median peak area of that metabolite within the same batch on the day the sample was run. The normalized peak area is then median scaled and imputed with the minimum across all samples. In this way, we can directly compare abundances relative to other samples for each metabolite. Relative abundance has no unit of measure. Finally we will identify interactions between prenatal vitamin D supplementation, rs12936231 genotype and sphingolipid metabolism in the risk of asthma/wheeze by age three. We will replicate this analysis in the COPSAC2010 population (ClinicalTrials.gov Identifier:NCT00856947).

VDAART Year 6 Analysis Plan

PRIMARY ANALYSIS: The null hypothesis of no treatment effect will be tested in a Cox Proportional Hazards Model of time to physician diagnosed asthma or onset of recurrent wheeze, adjusted for maternal levels of Vitamin D recorded at 10-18 weeks gestation, allowing for level by treatment interaction, and for any other relevant baseline covariates (race, maternal education, and clinical center), using the methods of Tsiatis et al. (Stat Med. 2008 October 15; 27(23): 4658-4677) to maximize precision of estimated treatment effect. The significance level for the test of no treatment effect will be 0.05.

SECONDARY ANALYSES: Effect estimates from all secondary analyses will be reported as point estimates with nominal 95% confidence intervals. Estimates will be derived from models adjusted for baseline maternal levels of Vitamin D as noted above.

Current active asthma, late onset recurrent wheeze, allergic sensitization, any allergic rhinitis, MD-diagnosed food allergy, food allergy with symptoms, eczema: Analysis is confined to individuals who provide data after age 5. Loss to followup is reasonably balanced between arms. Logistic regression will be used to test the hypothesis that there is no effect of treatment on risk of current active asthma. Separate tests will be conducted for no treatment effect on risk of late onset recurrent wheeze, on risk of allergic sensitization defined using specific IgE greater than or equal to 0.35IU, and on risk of allergic rhinitis birth to age 6. Similar models will be used separately to assess treatment effect on risk of eczema, active eczema, and food allergies.

Lower respiratory infections: The count of LRI per unit time will be modeled using negative binomial regression with covariates including treatment arm.

Impulse oscillometry: Analysis of treatment effect on impulse oscillometry components will be based on data available for 6 year old children, and will use linear modeling with adjustment for maternal baseline Vitamin D. A secondary analysis will examine treatment effect on trends in these measures through ages 4-6. This test will be based on mixed effects modeling.

Spirometry: Spirometric outcomes will be analyzed using linear models with transformations as needed, adjusting for race, age, sex and height. Bronchodilator response will be dichotomized at 10% of pre-challenge values, analyzed with logistic regression.

VDAART Asthma and/or Recurrent Wheeze Definitions for Primary Analysis (Time-to-Event)

Physician-diagnosed asthma Report of physician-diagnosed asthma at any time in the first 6 years of life. The time of onset will be the first report of wheeze OR the first report of use of asthma medication.

Recurrent wheeze - no diagnosis of asthma Caregiver report of wheeze OR use of any asthma medication on two separate years over the first 6 years. The time of onset will be the first report of wheeze OR the first report of use of asthma medication.

VDAART Year 6 Analyses - Definitions for Secondary Outcomes

Current Active Asthma Report of physician-diagnosed asthma at any time in the first 6 years of life, PLUS after the 5th birthday a) report of child's use of any asthma medication (see below) OR b) report of wheeze.

Recurrent Wheeze at age 6 yrs - no diagnosis of asthma At least 1 caregiver report of wheeze OR use of any asthma medication prior to the 3rd birthday, PLUS a report of wheeze OR use of any asthma medication after the 3rd birthday.

Late onset Recurrent wheeze - no diagnosis of asthma, wheeze, or asthma medication use prior to 3rd birthday A report of wheezing OR use of any asthma medication after the 5th birthday PLUS either wheezing or use of any asthma medication after the 3rd birthday but before the 5th birthday (between 3yrs and 5 yrs).

Total and specific IgE. Total and specific serum IgE will be measured year 6 samples from the children.

1. Total IgE will be analyzed as a continuous outcome.
2. Sensitization will be defined as any specific IgE ≥ 0.35 IU to the panel of allergens.

Allergic Rhinitis. This will be a positive response to the question "Since the last time we talked has a health care provider said that [CHILD] has hay fever, allergic rhinitis, or allergies involving the eyes or nose?" Any positive response from birth through age 6.

Eczema.

1. Ever eczema - positive response to "…has a health care provider said that [CHILD] has eczema?" at any time from birth through age 6.
2. Persistent eczema. Ever eczema at any time in the 6 years plus positive response to "itchy rash which was coming and going but did not completely get better?" after the 3rd birthday.

Lower Respiratory Infections (LRI). Lower respiratory tract infections (LRIs) will be defined based on caregiver responses to questionnaires. LRIs will be defined as a caregiver report of a physician's diagnosis of pneumonia, bronchiolitis, bronchitis, or croup (laryngotracheobronchitis). LRIs may occur multiple times over a six-year period in a child. Information on repeated episodes of LRI will be employed for rate estimation and comparison.

Food Allergies.

1. Doctor-diagnosis - any positive response from birth through age 6 to the question "In the last year, has a health care provider said that [CHILD] has food allergies?
2. Food allergy with symptoms - Doctor-diagnosis of food allergy PLUS any reaction to specific foods from the grid.

Lung Function.

1. Impulse oscillometry: R5, R20, AX, X5, R5-20, and R5-20% These variables will be used as continuous variables. The variables are measured at 4, 5, and 6 years of age. The primary analysis will look at values at 6 yrs of age, and a secondary analysis will investigate the trajectory (longitudinal analysis) from age 4 through 6 yrs.
2. Spirometry: pre- and post-bronchodilator FEV1, FVC, FEV1/FVC; Bronchodilator Response (BDR**). Analyses will adjust for race, age, sex, and height.

   * Asthma medication: rescue (inhaled beta-agonists or systemic corticosteroids) or controller medication (inhaled corticosteroids monotherapy, ICS/Long-acting beta-agonists, or leukotriene modifiers) ** A positive BDR will be defined as a change of 10% from the baseline FEV1 after inhalation of albuterol

ELIGIBILITY:
Inclusion Criteria:

* Personal history of asthma, eczema, allergic rhinitis or a history of asthma, eczema, allergic rhinitis in the biological father of the child
* Gestational age between 10 and 18 weeks at the time of randomization
* Maternal age between 18 and 39 years
* Not a current smoker
* English or Spanish speaking
* Intent to participate for the full 4 years (through Pregnancy and then until the 3rd birthday of the child)

Exclusion Criteria:

* Not meeting inclusion criteria
* Gestational age greater than 18 weeks
* Presence of chronic medical conditions
* Taking vitamin D supplements containing more than 2000 IU/day of vitamin D3
* Multiple gestation pregnancy (twins, triplets)
* Pregnancy achieved by assisted reproduction techniques (e.g., IUI, IVF)

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 876 (Actual)
Dates: Start 2009-09; Primary Completion 2015-01-21 (Actual); Study Completion 2023-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott T Weiss, Principal Investigator — Brigham and Women's Hospital
Locations (3):
- United States (3):
  - Robert Zeiger, MD, San Diego, California
  - George O'Connor, MD, Boston, Massachusetts
  - Leonard Bacharier, MD, St Louis, Missouri

REFERENCES:
- [Derived] Jung C, Lu Z, Litonjua AA, Loscalzo J, Weiss ST, Mirzakhani H. The association of early pregnancy vitamin D and BMI status with composite adverse pregnancy outcomes: an ancillary analysis of the Vitamin D Antenatal Asthma Reduction Trial. Am J Clin Nutr. 2025 Jul;122(1):324-334. doi: 10.1016/j.ajcnut.2025.04.034. Epub 2025 May 5. PMID 40334749
- [Derived] Kim M, Brustad N, Eliasen AU, Ali M, Wang T, Rasmussen MA, Ernst M, Hougaard D, Litonjua AA, Wheelock CE, Kelly RS, Chen Y, Prince N, Townsend PA, Stokholm J, Weiss ST, Bonnelykke K, Lasky-Su J, Chawes B. Bilirubin metabolism in early life and respiratory health during preschool age: A combined analysis of two independent birth cohorts. Med. 2024 Dec 13;5(12):1485-1494.e3. doi: 10.1016/j.medj.2024.07.021. Epub 2024 Aug 15. PMID 39151420
- [Derived] Palacios C, Kostiuk LL, Cuthbert A, Weeks J. Vitamin D supplementation for women during pregnancy. Cochrane Database Syst Rev. 2024 Jul 30;7(7):CD008873. doi: 10.1002/14651858.CD008873.pub5. PMID 39077939
- [Derived] Kim M, Brustad N, Ali M, Gurdeniz G, Arendt M, Litonjua AA, Wheelock CE, Kelly RS, Chen Y, Prince N, Guo F, Zhou X, Stokholm J, Bonnelykke K, Weiss ST, Bisgaard H, Lasky-Su J, Chawes B. Maternal vitamin D-related metabolome and offspring risk of asthma outcomes. J Allergy Clin Immunol. 2023 Dec;152(6):1646-1657.e11. doi: 10.1016/j.jaci.2023.06.030. Epub 2023 Aug 8. PMID 37558060
- [Derived] Prince N, Kelly RS, Chu SH, Kachroo P, Chen Y, Mendez KM, Begum S, Bisgaard H, Bonnelykke K, Kim M, Levy O, Litonjua AA, Wheelock CE, Weiss ST, Chawes BL, Lasky-Su JA. Elevated third trimester corticosteroid levels are associated with fewer offspring infections. Sci Rep. 2023 Jun 28;13(1):10461. doi: 10.1038/s41598-023-36535-0. PMID 37380711
- [Derived] Knihtila HM, Huang M, Prince N, Stubbs BJ, Carey VJ, Laranjo N, Mirzakhani H, Zeiger RS, Bacharier LB, O'Connor GT, Litonjua AA, Weiss ST, Lasky-Su J. Maternal vitamin D status modifies the effects of early life tobacco exposure on child lung function. J Allergy Clin Immunol. 2023 Feb;151(2):556-564. doi: 10.1016/j.jaci.2022.10.030. Epub 2022 Nov 16. PMID 36400177
- [Derived] Lee-Sarwar KA, Chen YC, Chen YY, Kozyrskyj AL, Mandhane PJ, Turvey SE, Subbarao P, Bisgaard H, Stokholm J, Chawes B, Sorensen SJ, Kelly RS, Lasky-Su J, Zeiger RS, O'Connor GT, Sandel MT, Bacharier LB, Beigelman A, Carey VJ, Harshfield BJ, Laranjo N, Gold DR, Weiss ST, Litonjua AA. The maternal prenatal and offspring early-life gut microbiome of childhood asthma phenotypes. Allergy. 2023 Feb;78(2):418-428. doi: 10.1111/all.15516. Epub 2022 Sep 24. PMID 36107703
- [Derived] Knihtila HM, Kelly RS, Brustad N, Huang M, Kachroo P, Chawes BL, Stokholm J, Bonnelykke K, Pedersen CT, Bisgaard H, Litonjua AA, Lasky-Su JA, Weiss ST. Maternal 17q21 genotype influences prenatal vitamin D effects on offspring asthma/recurrent wheeze. Eur Respir J. 2021 Sep 23;58(3):2002012. doi: 10.1183/13993003.02012-2020. Print 2021 Sep. PMID 33653805
- [Derived] Litonjua AA, Carey VJ, Laranjo N, Stubbs BJ, Mirzakhani H, O'Connor GT, Sandel M, Beigelman A, Bacharier LB, Zeiger RS, Schatz M, Hollis BW, Weiss ST. Six-Year Follow-up of a Trial of Antenatal Vitamin D for Asthma Reduction. N Engl J Med. 2020 Feb 6;382(6):525-533. doi: 10.1056/NEJMoa1906137. PMID 32023372
- [Derived] Lu M, Hollis BW, Carey VJ, Laranjo N, Singh RJ, Weiss ST, Litonjua AA. Determinants and Measurement of Neonatal Vitamin D: Overestimation of 25(OH)D in Cord Blood Using CLIA Assay Technology. J Clin Endocrinol Metab. 2020 Apr 1;105(4):e1085-92. doi: 10.1210/clinem/dgz299. PMID 31872219
- [Derived] Lee-Sarwar KA, Kelly RS, Lasky-Su J, Zeiger RS, O'Connor GT, Sandel MT, Bacharier LB, Beigelman A, Rifas-Shiman SL, Carey VJ, Harshfield BJ, Laranjo N, Gold DR, Weiss ST, Litonjua AA. Fecal short-chain fatty acids in pregnancy and offspring asthma and allergic outcomes. J Allergy Clin Immunol Pract. 2020 Mar;8(3):1100-1102.e13. doi: 10.1016/j.jaip.2019.08.036. Epub 2019 Sep 5. No abstract available. PMID 31494295
- [Derived] Yu B, Zanetti KA, Temprosa M, Albanes D, Appel N, Barrera CB, Ben-Shlomo Y, Boerwinkle E, Casas JP, Clish C, Dale C, Dehghan A, Derkach A, Eliassen AH, Elliott P, Fahy E, Gieger C, Gunter MJ, Harada S, Harris T, Herr DR, Herrington D, Hirschhorn JN, Hoover E, Hsing AW, Johansson M, Kelly RS, Khoo CM, Kivimaki M, Kristal BS, Langenberg C, Lasky-Su J, Lawlor DA, Lotta LA, Mangino M, Le Marchand L, Mathe E, Matthews CE, Menni C, Mucci LA, Murphy R, Oresic M, Orwoll E, Ose J, Pereira AC, Playdon MC, Poston L, Price J, Qi Q, Rexrode K, Risch A, Sampson J, Seow WJ, Sesso HD, Shah SH, Shu XO, Smith GCS, Sovio U, Stevens VL, Stolzenberg-Solomon R, Takebayashi T, Tillin T, Travis R, Tzoulaki I, Ulrich CM, Vasan RS, Verma M, Wang Y, Wareham NJ, Wong A, Younes N, Zhao H, Zheng W, Moore SC. The Consortium of Metabolomics Studies (COMETS): Metabolomics in 47 Prospective Cohort Studies. Am J Epidemiol. 2019 Jun 1;188(6):991-1012. doi: 10.1093/aje/kwz028. PMID 31155658
- [Derived] Lee-Sarwar KA, Kelly RS, Lasky-Su J, Zeiger RS, O'Connor GT, Sandel MT, Bacharier LB, Beigelman A, Laranjo N, Gold DR, Weiss ST, Litonjua AA. Integrative analysis of the intestinal metabolome of childhood asthma. J Allergy Clin Immunol. 2019 Aug;144(2):442-454. doi: 10.1016/j.jaci.2019.02.032. Epub 2019 Mar 23. PMID 30914378
- [Derived] Mirzakhani H, Carey VJ, Zeiger R, Bacharier LB, O'Connor GT, Schatz MX, Laranjo N, Weiss ST, Litonjua AA. Impact of parental asthma, prenatal maternal asthma control, and vitamin D status on risk of asthma and recurrent wheeze in 3-year-old children. Clin Exp Allergy. 2019 Apr;49(4):419-429. doi: 10.1111/cea.13320. Epub 2019 Jan 3. PMID 30461089
- [Derived] Savage JH, Lee-Sarwar KA, Sordillo JE, Lange NE, Zhou Y, O'Connor GT, Sandel M, Bacharier LB, Zeiger R, Sodergren E, Weinstock GM, Gold DR, Weiss ST, Litonjua AA. Diet during Pregnancy and Infancy and the Infant Intestinal Microbiome. J Pediatr. 2018 Dec;203:47-54.e4. doi: 10.1016/j.jpeds.2018.07.066. Epub 2018 Aug 30. PMID 30173873
- [Derived] Mirzakhani H, Carey VJ, McElrath TF, Qiu W, Hollis BW, O'Connor GT, Zeiger RS, Bacharier L, Litonjua AA, Weiss ST. Impact of Preeclampsia on the Relationship between Maternal Asthma and Offspring Asthma. An Observation from the VDAART Clinical Trial. Am J Respir Crit Care Med. 2019 Jan 1;199(1):32-42. doi: 10.1164/rccm.201804-0770OC. PMID 30153046
- [Derived] Mirzakhani H, Al-Garawi AA, Carey VJ, Qiu W, Litonjua AA, Weiss ST. Expression network analysis reveals cord blood vitamin D-associated genes affecting risk of early life wheeze. Thorax. 2019 Feb;74(2):200-202. doi: 10.1136/thoraxjnl-2018-211962. Epub 2018 Jul 18. PMID 30021811
- [Derived] Kelly RS, Sordillo JE, Lasky-Su J, Dahlin A, Perng W, Rifas-Shiman SL, Weiss ST, Gold DR, Litonjua AA, Hivert MF, Oken E, Wu AC. Plasma metabolite profiles in children with current asthma. Clin Exp Allergy. 2018 Oct;48(10):1297-1304. doi: 10.1111/cea.13183. Epub 2018 Jul 3. PMID 29808611
- [Derived] Wolsk HM, Chawes BL, Litonjua AA, Hollis BW, Waage J, Stokholm J, Bonnelykke K, Bisgaard H, Weiss ST. Prenatal vitamin D supplementation reduces risk of asthma/recurrent wheeze in early childhood: A combined analysis of two randomized controlled trials. PLoS One. 2017 Oct 27;12(10):e0186657. doi: 10.1371/journal.pone.0186657. eCollection 2017. PMID 29077711
- [Derived] Blighe K, Chawes BL, Kelly RS, Mirzakhani H, McGeachie M, Litonjua AA, Weiss ST, Lasky-Su JA. Vitamin D prenatal programming of childhood metabolomics profiles at age 3 y. Am J Clin Nutr. 2017 Oct;106(4):1092-1099. doi: 10.3945/ajcn.117.158220. Epub 2017 Aug 23. PMID 28835366
- [Derived] Mirzakhani H, O'Connor G, Bacharier LB, Zeiger RS, Schatz MX, Weiss ST, Litonjua AA. Asthma control status in pregnancy, body mass index, and maternal vitamin D levels. J Allergy Clin Immunol. 2017 Nov;140(5):1453-1456.e7. doi: 10.1016/j.jaci.2017.03.053. Epub 2017 Jun 9. PMID 28606587
- [Derived] Hornsby E, Pfeffer PE, Laranjo N, Cruikshank W, Tuzova M, Litonjua AA, Weiss ST, Carey VJ, O'Connor G, Hawrylowicz C. Vitamin D supplementation during pregnancy: Effect on the neonatal immune system in a randomized controlled trial. J Allergy Clin Immunol. 2018 Jan;141(1):269-278.e1. doi: 10.1016/j.jaci.2017.02.039. Epub 2017 May 26. PMID 28552588
- [Derived] Mirzakhani H, Litonjua AA, McElrath TF, O'Connor G, Lee-Parritz A, Iverson R, Macones G, Strunk RC, Bacharier LB, Zeiger R, Hollis BW, Handy DE, Sharma A, Laranjo N, Carey V, Qiu W, Santolini M, Liu S, Chhabra D, Enquobahrie DA, Williams MA, Loscalzo J, Weiss ST. Early pregnancy vitamin D status and risk of preeclampsia. J Clin Invest. 2016 Dec 1;126(12):4702-4715. doi: 10.1172/JCI89031. Epub 2016 Nov 14. PMID 27841759
- [Derived] Al-Garawi A, Carey VJ, Chhabra D, Mirzakhani H, Morrow J, Lasky-Su J, Qiu W, Laranjo N, Litonjua AA, Weiss ST. The Role of Vitamin D in the Transcriptional Program of Human Pregnancy. PLoS One. 2016 Oct 6;11(10):e0163832. doi: 10.1371/journal.pone.0163832. eCollection 2016. PMID 27711190
- [Derived] Litonjua AA, Carey VJ, Laranjo N, Harshfield BJ, McElrath TF, O'Connor GT, Sandel M, Iverson RE Jr, Lee-Paritz A, Strunk RC, Bacharier LB, Macones GA, Zeiger RS, Schatz M, Hollis BW, Hornsby E, Hawrylowicz C, Wu AC, Weiss ST. Effect of Prenatal Supplementation With Vitamin D on Asthma or Recurrent Wheezing in Offspring by Age 3 Years: The VDAART Randomized Clinical Trial. JAMA. 2016 Jan 26;315(4):362-70. doi: 10.1001/jama.2015.18589. PMID 26813209

RESULTS

PARTICIPANT FLOW:
Recruitment Details: VDAART was a randomized, double-blind, placebo-controlled trial. Enrollment began October 2009 and completed follow-up January 2015 in 3 medical centers in the United Stated. 881 pregnant women age 18-39 at high risk for having children with asthma were randomized at 10-18 weeks gestation. 5 did not meet inclusion criteria and were removed.
Groups:
- Vitamin D Treatment (Mothers): Mothers' assigned to vitamin D (daily 4,000 IU vitamin D plus a multivitamin with 400 IU vitamin D).
- Placebo (Mothers): Mothers' assigned to placebo (daily placebo pill plus a multivitamin with 400 IU vitamin D). Serves as the "Control" (providing the current standard of care during pregnancy).
- Vitamin D Treatment (Offspring): Offspring of mothers' assigned to vitamin D (daily 4,000 IU vitamin D plus a multivitamin with 400 IU vitamin D)
- Placebo (Offspring): Offspring of mothers' assigned to placebo (daily placebo pill plus a multivitamin with 400 IU vitamin D). Serves as the "Control"
Period: Overall Study
Arm/Group | Vitamin D Treatment (Mothers) | Placebo (Mothers) | Vitamin D Treatment (Offspring) | Placebo (Offspring)
Started | 440 | 436 | 440 | 436
Completed | 386 | 391 | 405 | 401
Not Completed | 54 | 45 | 35 | 35
Not completed — Lost to Follow-up | 16 | 17 | 19 | 21
Not completed — Fetal/neonatal deaths | 16 | 14 | 16 | 14
Not completed — Blood sample not collected | 22 | 14 | 0 | 0

BASELINE CHARACTERISTICS:
Population: For the treatment arm, 440 were randomized. For the placebo/control arm, 436 were randomized. Some mothers dropped out of the study, prior to delivery. And not all of the pregnancies resulted in a live birth, hence the differences between the 440 mothers and 405 children on the treatment arm and 436 mothers and 401 children on the control arm.
Groups:
- Vitamin D Treatment (Children): Children of mothers' assigned to vitamin D (daily 4,000 IU vitamin D plus a multivitamin with 400 IU vitamin D).
- Placebo (Children): Children of mothers' assigned to placebo (daily placebo pill plus a multivitamin with 400 IU vitamin D). Serves as the "Control" (providing the current standard of care during pregnancy).
- Total: Total of all reporting groups
Arm/Group | Vitamin D Treatment (Mothers) | Placebo (Mothers) | Vitamin D Treatment (Children) | Placebo (Children) | Total
Number analyzed (Participants) | 440 | 436 | 405 | 401 | 1682
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (5.5) | 27.3 (5.6) | 0 (0) | 0 (0) | 27.4 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 440 | 436 | 204 | 181 | 1261
  Male | 0 | 0 | 201 | 220 | 421
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 190 | 190 | 199 | 191 | 770
  White Hispanic | 59 | 61 | 53 | 51 | 224
  White non-Hispanic | 114 | 116 | 82 | 79 | 391
  Other | 77 | 69 | 71 | 80 | 297

OUTCOME MEASURES:

1. Primary Outcome: Asthma or Recurrent Wheeze in First 3 Years of Life
Description: Parental report of physician diagnosis of asthma or occurrence of recurrent wheeze in the child's first 3 years of life ascertained from questionnaires administered every 3 months.
  *For some variables the "negative" count incorporates "negative and indeterminate."
Time Frame: First 3 years of life.
Population: Some measures have missing data due to collection, technical, and processing issues.
Measure: Count of Participants; unit: Participants
Groups:
- Vitamin D Treatment: Children of mother's assigned 4400 IU Vitamin D
- Placebo: Children of mother's assigned 400 IU Vitamin D.
Arm/Group | Vitamin D Treatment | Placebo
Number analyzed (Participants) | 405 | 401
Participants
  Children positive | 98 | 120
  Children negative | 307 | 281

2. Primary Outcome: Achieved Maternal 25(OH)D Level of ≥ 30 ng/mL at Third Trimester Sampling.
Description: Maternal serum 25-hydroxyvitamin D measurement at third trimester during pregnancy
Time Frame: 32-38 weeks gestation
Population: Some measures have missing data due to collection, technical, and processing issues.
Measure: Count of Participants; unit: Participants
Groups:
- Vitamin D Treatment: Mothers' assigned to vitamin D (daily 4,000 IU vitamin D plus a multivitamin with 400 IU vitamin D).
- Placebo: Mothers' assigned to placebo (daily placebo pill plus a multivitamin with 400 IU vitamin D). Serves as the "Control" (providing the current standard of care during pregnancy).
Arm/Group | Vitamin D Treatment | Placebo
Number analyzed (Participants) | 386 | 391
Participants
  25(OH)D level of ≥ 30 ng/mL , women positive | 289 | 133
  25(OH)D level of ≥ 30 ng/mL , women negative | 97 | 258

3. Secondary Outcome: Child Positive-specific IgE Tests From Blood Collection at 3 Year Visit.
Description: Child positive-specific IgE tests from blood collection at 3 year visit.
Time Frame: 3 years
Population: Some measures have missing data due to collection, technical, and processing issues.
Measure: Number; unit: Positive-specific IgE tests
Units Other Than Participants: completed tests
Arm/Group | Vitamin D Treatment | Placebo
Number analyzed (Participants) | 278 | 263
Number analyzed (completed tests) | 3876 | 3651
Positive-specific IgE tests | 414 | 452

4. Secondary Outcome: Child Serum 25-hydroxyvitamin D Measurement From Blood Collection at 1 Year Visit.
Description: Child serum 25-hydroxyvitamin D measurement from blood collection at 1 year visit.
Time Frame: 1 year visit
Population: Some measures have missing data due to collection, technical, and processing issues.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vitamin D Treatment | Placebo
Number analyzed (Participants) | 322 | 309
ng/mL | 29.3 (9.2) | 30.1 (10.8)

5. Secondary Outcome: Parental Report of Physician Diagnosed Eczema (With Rash) in the Child's First 3 Years of Life.
Description: Parental report of physician diagnosis of eczema with rash in typical distribution in the child's first 3 years of life ascertained from questionnaires administered every 3 months.
  *For some variables the "negative" count incorporates "negative and indeterminate."
Time Frame: Child's first 3 years of life.
Population: Some measures have missing data due to collection, technical, and processing issues.
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D Treatment | Placebo
Number analyzed (Participants) | 405 | 401
Participants
  Children positive | 83 | 89
  Children negative | 322 | 312

6. Secondary Outcome: Parental Report of Physician Diagnosis of Lower Respiratory Tract Infection in the Child's First 3 Years of Life.
Description: Parental report of physician diagnosis of lower respiratory tract infection (LRI) in the child's first 3 years of life. LRI defined as physician diagnosed bronchitis, bronchiolitis, croup, or pneumonia ascertained from questionnaires administered every 3 months.
Time Frame: Child's first 3 years of life.
Population: Some measures have missing data due to collection, technical, and processing issues.
Measure: Number; unit: Number of lower respiratory infections
Arm/Group | Vitamin D Treatment | Placebo
Number analyzed (Participants) | 405 | 401
Number of lower respiratory infections | 222 | 276

7. Secondary Outcome: Child Serum 25-hydroxyvitamin D Measurement From Blood Collection at 3 Year Visit.
Description: Child serum 25-hydroxyvitamin D measurement from blood collection at 3 year visit.
Time Frame: Blood collection at childs' 3 year visit.
Population: Some measures have missing data due to collection, technical, and processing issues.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vitamin D Treatment | Placebo
Number analyzed (Participants) | 289 | 271
ng/mL | 21.3 (10.4) | 21.5 (8.5)

8. Secondary Outcome: Any Allergic Sensitization in the Child's First 3 Years of Life.
Description: Any allergic sensitization in the child's first 3 years of life.
  *For some variables the "negative" count incorporates "negative and indeterminate."
Time Frame: Child's first 3 years of life.
Population: Some measures have missing data due to collection, technical, and processing issues.
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D Treatment | Placebo
Number analyzed (Participants) | 278 | 261
Participants
  Any sensitization | 146 | 144
  No sensitization | 132 | 117

9. Secondary Outcome: Mass Spec Vitamin D Value From Cord Blood at Delivery
Description: Mass Spec Vitamin D value from cord blood at delivery
Time Frame: Blood collection at delivery
Population: Some measures have missing data due to collection, technical, and processing issues.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vitamin D Treatment | Placebo
Number analyzed (Participants) | 303 | 316
ng/mL | 28.2 (12.4) | 19.1 (9.7)

10. Secondary Outcome: Sphingolipid Profile
Description: Mass spec measured relative abundance of five metabolites of the sphingolipid metabolism pathway in plasma samples extracted at the year one visit.
Time Frame: 1 year
Population: Some measures have missing data due to collection, technical, and processing issues.
Measure: Mean (Standard Deviation); unit: relative abundance (no units)
Arm/Group | Vitamin D Treatment | Placebo
Number analyzed (Participants) | 211 | 202
relative abundance (no units)
  sphinganine-1-phosphate | 0.32 (0.10) | 0.32 (0.10)
  sphinganine | 0.33 (0.20) | 0.31 (0.18)
  phosphoethanolamine | 0.33 (0.13) | 0.34 (0.13)
  sphingosine | 0.34 (0.17) | 0.33 (0.17)
  sphingosine-1-phosphate | 0.31 (0.06) | 0.32 (0.06)

11. Secondary Outcome: Sphingolipid Profile
Description: Mass spec measured relative abundance of five metabolites of the sphingolipid metabolism pathway in plasma samples extracted at the year three visit.
Time Frame: 3 years
Population: Some measures have missing data due to collection, technical, and processing issues.
Measure: Mean (Standard Deviation); unit: relative abundance (no units)
Arm/Group | Vitamin D Treatment | Placebo
Number analyzed (Participants) | 179 | 174
relative abundance (no units)
  sphinganine-1-phosphate | 0.34 (0.12) | 0.32 (0.12)
  sphinganine | 0.39 (0.20) | 0.37 (0.20)
  phosphoethanolamine | 0.31 (0.11) | 0.30 (0.11)
  sphingosine | 0.38 (0.19) | 0.37 (0.19)
  sphingosine-1-phosphate | 0.31 (0.07) | 0.30 (0.08)

12. Secondary Outcome: Child 17q21 Genotype
Description: Genotype at the rs12936231 SNP
Time Frame: 3 years
Population: Some measures have missing data due to collection, technical, and processing issues.
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D Treatment | Placebo
Number analyzed (Participants) | 311 | 307
Participants
  CC | 93 | 78
  GC | 152 | 161
  GG | 66 | 68

13. Secondary Outcome: Fecal Microbiome Profile
Description: We extracted DNA and sequenced the bacterial 16S V4 hyper-variable region. The average number of 16S region reads sequenced per participant is provided here. Prior evidence suggests that read counts of at least 1,000 are adequate for 16S fecal microbiome profiling (Reference: Momozawa Y, et cal. Characterization of bacteria in biopsies of colon and stools by high throughput sequencing of the V2 region of bacterial 16S rRNA gene in human. PLoS One. 2011 Feb 10;6(2):e16952.)
Time Frame: Mother at 32-38 weeks gestation, Child's first 6 years of life
Measure: Mean (Standard Deviation); unit: read counts
Units Other Than Participants: Samples
Arm/Group | Vitamin D Treatment | Placebo
Number analyzed (Participants) | 335 | 332
Number analyzed (Samples) | 696 | 631
read counts
  Mother at 32-38 weeks gestation | 10787 (3534) | 10773 (2511)
  Child at 3-6 months | 13443 (8624) | 14024 (9010)
  Child at 1 year | 11709 (4202) | 11635 (3488)
  Child at 3 years | 12095 (4733) | 12407 (4288)
  Child at 4 years | 0 (0) | 0 (0)
  Child at 5 years | 0 (0) | 0 (0)
  Child at 6 years | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: From the point mothers entered the study until 2 years post delivery.
Description: Maternal and offspring SAEs were collected via a monthly electronic record review and via quarterly follow-up calls.
Groups:
- Placebo (Offspring): Offspring of mothers' assigned to placebo (daily placebo pill plus a multivitamin with 400 IU vitamin D). Serves as the "Control" (providing the current standard of care during pregnancy).
Arm/Group | Vitamin D Treatment (Mothers) | Placebo (Mothers) | Vitamin D Treatment (Offspring) | Placebo (Offspring)
All-Cause Mortality (participants affected / at risk) | 0/440 | 1/436 | 3/440 | 3/436
Serious Adverse Events (participants affected / at risk) | 75/440 | 77/436 | 58/440 | 52/436
Other Adverse Events (participants affected / at risk) | 0/440 | 0/436 | 0/440 | 0/436
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D Treatment (Mothers) (N=440) | Placebo (Mothers) (N=436) | Vitamin D Treatment (Offspring) (N=440) | Placebo (Offspring) (N=436)
HELLP (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 34 (36) | 37 (38) | 0 (0) | 0 (0)
Hospitalization (General disorders) | 32 (42) | 32 (45) | 0 (0) | 0 (0)
Postpartum Hospitalization (General disorders) | 7 (10) | 6 (8) | 0 (0) | 0 (0)
Pre-term delivery <32 weeks gestation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 3 (5) | 7 (11)
Maternal Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major fetal or congenital anomaly (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 10 (17) | 13 (14)
NICU (General disorders) | 0 (0) | 0 (0) | 29 (36) | 18 (28) — Neonatal ICU admission
Still birth or intrauterine fetal death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 13 (13) | 11 (11)
Neonatal demise (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No